CLINICAL TRIAL: NCT00633321
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Multicenter, Dose-Ranging Study of 100 or 250 μg of TA-NIC to Assess the Efficacy and Safety of the Vaccine as an Aid to Smoking Cessation
Brief Title: Study of TA-NIC to Assess the Efficacy and Safety of the Vaccine as an Aid to Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celtic Pharma Development Services (Industry)
Responsible Party: Patrick O'Connor, MD, PhD - Head of Clinical Developement, Celtic Pharmaceutical Developement
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TA-NIC/04
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Smoking
Keywords: smoking cessation; quit smoking; smoking vaccine; nicotine vaccine; TA-NIC; Aid for smoking cessation in smokers motivated to quit
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — TA-NIC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): TA-NIC 100 μg
  Interventions: Biological: TA-NIC
- 2 (Experimental): TA-NIC 250 μg
  Interventions: Biological: TA-NIC
- 3 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TA-NIC — TA-NIC vaccine will be administered to each subject as 7 single doses administered at Weeks 0, 2, 4, 6, 8, 12, and 16.
  Arms: 1; 2
Biological: Placebo — Placebo will be administered to each subject as 7 single doses administered at Weeks 0, 2, 4, 6, 8, 12, and 16.
  Arms: 3

SUMMARY:
Over 1 billion people worldwide smoke, resulting in an estimated 4 million deaths annually from smoking-related disease.1 Persistent and long-term smoking leads to an increased risk of cardiovascular damage, respiratory disease, and a higher incidence of a variety of cancers; but for smokers who can quit there is an immediate and significant beneficial impact on their health and life expectancy. Cigarette smoking remains the leading preventable cause of death in the United States (US), accounting for approximately 1 of every 5 deaths (438,000 people) each year.

This Phase 2 study will investigate the efficacy and tolerability of 2 doses of TA-NIC compared to placebo as an aid to smoking cessation in smokers who are motivated to quit.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebocontrolled, 3-arm, Phase 2 study evaluating the efficacy and safety of TA-NIC as an aid for smoking cessation in smokers motivated to quit within 12 weeks. At the start of the study, each subject will set a Target Quit Date, which must be within 12 weeks after first injection. Each subject will receive 7 injections (vaccinations) from Weeks 0 to 16. Subjects will be encouraged to follow a phased reduction in cigarette consumption leading up to the Target Quit Date. All vaccinated subjects will be offered a counseling session at each clinic visit and will be contacted by telephone at Weeks 1, 3, 5, 7, 9, 14, 18, and 21 to provide up to 10 minutes of support and counseling for their smoking cessation. Smoking cessation will be measured during a 4-week assessment period from Week 22 to Week 26. Smoking cessation will be defined as complete abstinence during this 4-week period. Subject follow-up will continue to Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Female subjects must be either of non child bearing potential (i.e., either surgically sterilized or post menopausal) or must be using adequate contraception, have a negative pregnancy test and must agree to continue to use such precautions for 3 months after the last immunization. Acceptable contraceptive methods are oral or parenteral hormonal contraceptives; intrauterine device; barrier and spermicide. Abstinence or partner vasectomy are not acceptable methods.
* A "smoker" who has smoked on a regular basis for a least a year and is currently smoking at least 10 cigarettes per day
* Is motivated to quit smoking in the next 12 weeks
* Agrees to avoid smoking cessation pharmacotherapies, and any other methods of smoking cessation, other than those provided as part of this protocol
* Has good general health as determined by medical history, general clinical examination, vital signs (systolic blood pressure ≤140 mm Hg, diastolic blood pressure ≤90 mm Hg, heart rate ≤100 beats per minute, and body temperature of 36.1°-37.8° C), and clinical laboratory test results; and has a World Health Organization (WHO) performance status of 0 or 1 (see Appendix A for WHO performance status scale)
* Has provided written informed consent.

Exclusion Criteria:

* Have known immunodeficiency, or tested positive for human immunodeficiency virus (HIV) or hepatitis B at screening.
* Are taking medication known to have significant immunosuppressive effects such as systemic glucocorticoids (topical and inhaled formulations are permitted)
* Are intending to use other forms of smoking cessation pharmacotherapies or other methods of smoking cessation during the period of the study, other than those provided as part of this protocol; or who are receiving smoking cessation products (e.g., bupropion, clonidine, nortriptyline) for indications other than smoking cessation during the period of study
* History of sensitivity to aluminum hydroxide gel
* History of severe adverse reaction to cholera vaccine
* Known current user of drugs of abuse, or with a recent history (within the past 6 months) of use of drugs of abuse
* Recent (within the past 6 months) history of alcohol abuse
* Current non-cigarette tobacco use
* Previous vaccination with TA-NIC
* Participation in another clinical study within 30 days before study entry
* Female subjects with a positive pregnancy test; lactating mothers; women of child-bearing potential who do not agree to continue adequate contraception (i.e., oral or parenteral hormonal contraceptives, intrauterine device, barrier, and/or spermicide) and pregnancy tests from start of study through 3 months after the last immunization; or women who are planning to become pregnant during the period of the study
* Clinical laboratory value outside the normal range of the central laboratory (see Appendix G), unless the value has been justified by the Investigator in writing
* Any other factor that in the opinion of the Investigator would make the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
4-week assessment period quit rate at Week 26 measured by self-reported abstinence in the 4 weeks immediately prior to the 26 week visit and supported by CO breath test data | Week 26

SECONDARY OUTCOMES:
Measures of anti-nicotine antibody levels at key study visits | Prospective
Quit status at the final follow-up visit (Week 52) | Week 52
CO breath test measurements at key study visits | Prospective
Serum cotinine levels at key study visits | Prospective
Nicotine dependence as measured by Fagerström score, for those subjects who are still smokers | Prospective
Urge to smoke (craving) and smoking satisfaction, as measured by QSU-brief and mCEQ, respectively | Prospective
Continuous abstinence between Weeks 26 and 52 | Prospective
Safety and tolerability of TA-NIC | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Krefetz, Principal Investigator — CNS Research Institute, P.C; Gruener, Principal Investigator — CRI Worldwide, LLC; Coats, Principal Investigator — Benchmark Research; Rarick, Principal Investigator — Benchmark Research; Seger, Principal Investigator — Benchmark Research - Fort Worth; Jeanfreau, Principal Investigator — Benchmark Research; Geller, Principal Investigator — Centennial Medical Group; Saway, Principal Investigator — Columbia Medical Practice; Dale, Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - Benchmark Research, Sacramento, California
  - Benchmark Research, Metairie, Louisiana
  - Columbia Medical Practice, Columbia, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - CNS Research Institute, P.C., Clementon, New Jersey
  - CRI Worldwide, LLC Kirkbride Center, Philadelphia, Pennsylvania
  - Benchmark Research, Austin, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas

REFERENCES:
- [Background] Doll R, Hill AB. The mortality of doctors in relation to their smoking habits: a preliminary report. 1954. BMJ. 2004 Jun 26;328(7455):1529-33; discussion 1533. doi: 10.1136/bmj.328.7455.1529. No abstract available. PMID 15217868
- [Background] Centers for Disease Control and Prevention (CDC). Annual smoking-attributable mortality, years of potential life lost, and economic costs--United States, 1995-1999. MMWR Morb Mortal Wkly Rep. 2002 Apr 12;51(14):300-3. PMID 12002168
- [Background] Centers for Disease Control and Prevention (CDC). Annual smoking-attributable mortality, years of potential life lost, and productivity losses--United States, 1997-2001. MMWR Morb Mortal Wkly Rep. 2005 Jul 1;54(25):625-8. PMID 15988406
- [Background] Silagy C, Lancaster T, Stead L, Mant D, Fowler G. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2004;(3):CD000146. doi: 10.1002/14651858.CD000146.pub2. PMID 15266423
- [Background] Hall SM, Humfleet GL, Reus VI, Munoz RF, Hartz DT, Maude-Griffin R. Psychological intervention and antidepressant treatment in smoking cessation. Arch Gen Psychiatry. 2002 Oct;59(10):930-6. doi: 10.1001/archpsyc.59.10.930. PMID 12365880
- [Background] Hughes JR, Stead LF, Lancaster T. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD000031. doi: 10.1002/14651858.CD000031.pub3. PMID 17253443
- [Background] Jorenby DE, Leischow SJ, Nides MA, Rennard SI, Johnston JA, Hughes AR, Smith SS, Muramoto ML, Daughton DM, Doan K, Fiore MC, Baker TB. A controlled trial of sustained-release bupropion, a nicotine patch, or both for smoking cessation. N Engl J Med. 1999 Mar 4;340(9):685-91. doi: 10.1056/NEJM199903043400903. PMID 10053177
- [Background] Silagy C, Mant D, Fowler G, Lodge M. Meta-analysis on efficacy of nicotine replacement therapies in smoking cessation. Lancet. 1994 Jan 15;343(8890):139-42. doi: 10.1016/s0140-6736(94)90933-4. PMID 7904003
- [Background] West RJ, Russell MA. Cardiovascular and subjective effects of smoking before and after 24 h of abstinence from cigarettes. Psychopharmacology (Berl). 1987;92(1):118-21. doi: 10.1007/BF00215491. PMID 3110822
- [Background] Pentel PR, Malin DH, Ennifar S, Hieda Y, Keyler DE, Lake JR, Milstein JR, Basham LE, Coy RT, Moon JW, Naso R, Fattom A. A nicotine conjugate vaccine reduces nicotine distribution to brain and attenuates its behavioral and cardiovascular effects in rats. Pharmacol Biochem Behav. 2000 Jan 1;65(1):191-8. doi: 10.1016/s0091-3057(99)00206-3. PMID 10638653
- [Background] Malin DH, Lake JR, Lin A, Saldana M, Balch L, Irvin ML, Chandrasekara H, Alvarado CL, Hieda Y, Keyler DE, Pentel PR, Ennifar S, Basham LE, Naso R, Fattom A. Passive immunization against nicotine prevents nicotine alleviation of nicotine abstinence syndrome. Pharmacol Biochem Behav. 2001 Jan;68(1):87-92. doi: 10.1016/s0091-3057(00)00436-6. PMID 11274712
- [Background] Hieda Y, Keyler DE, VanDeVoort JT, Niedbala RS, Raphael DE, Ross CA, Pentel PR. Immunization of rats reduces nicotine distribution to brain. Psychopharmacology (Berl). 1999 Apr;143(2):150-7. doi: 10.1007/s002130050930. PMID 10326777
- [Background] Hieda Y, Keyler DE, Ennifar S, Fattom A, Pentel PR. Vaccination against nicotine during continued nicotine administration in rats: immunogenicity of the vaccine and effects on nicotine distribution to brain. Int J Immunopharmacol. 2000 Oct;22(10):809-19. doi: 10.1016/s0192-0561(00)00042-4. PMID 10963853
- [Background] Fagerstrom KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire. J Behav Med. 1989 Apr;12(2):159-82. doi: 10.1007/BF00846549. PMID 2668531
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Kozlowski LT, Porter CQ, Orleans CT, Pope MA, Heatherton T. Predicting smoking cessation with self-reported measures of nicotine dependence: FTQ, FTND, and HSI. Drug Alcohol Depend. 1994 Feb;34(3):211-6. doi: 10.1016/0376-8716(94)90158-9. PMID 8033758
- [Background] Hurt RD, Sachs DP, Glover ED, Offord KP, Johnston JA, Dale LC, Khayrallah MA, Schroeder DR, Glover PN, Sullivan CR, Croghan IT, Sullivan PM. A comparison of sustained-release bupropion and placebo for smoking cessation. N Engl J Med. 1997 Oct 23;337(17):1195-202. doi: 10.1056/NEJM199710233371703. PMID 9337378
- [Background] Hays JT, Hurt RD, Rigotti NA, Niaura R, Gonzales D, Durcan MJ, Sachs DP, Wolter TD, Buist AS, Johnston JA, White JD. Sustained-release bupropion for pharmacologic relapse prevention after smoking cessation. a randomized, controlled trial. Ann Intern Med. 2001 Sep 18;135(6):423-33. doi: 10.7326/0003-4819-135-6-200109180-00011. PMID 11560455
- [Background] Brauer LH, Behm FM, Lane JD, Westman EC, Perkins C, Rose JE. Individual differences in smoking reward from de-nicotinized cigarettes. Nicotine Tob Res. 2001 May;3(2):101-9. doi: 10.1080/14622200123249. PMID 11403723
- [Background] Rose JE, Behm FM, Westman EC, Levin ED, Stein RM, Ripka GV. Mecamylamine combined with nicotine skin patch facilitates smoking cessation beyond nicotine patch treatment alone. Clin Pharmacol Ther. 1994 Jul;56(1):86-99. doi: 10.1038/clpt.1994.105. PMID 8033499
- [Background] Rose JE, Behm FM, Westman EC. Nicotine-mecamylamine treatment for smoking cessation: the role of pre-cessation therapy. Exp Clin Psychopharmacol. 1998 Aug;6(3):331-43. doi: 10.1037//1064-1297.6.3.331. PMID 9725117
- [Background] Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Confirmatory factor analyses and reliability of the modified cigarette evaluation questionnaire. Addict Behav. 2007 May;32(5):912-23. doi: 10.1016/j.addbeh.2006.06.028. Epub 2006 Jul 27. PMID 16875787
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] World Health Organization; Tobacco Free Initiative: Why is tobacco a public health priority? http:www.who.int/tobacco/en
- [Background] Fiore MC, Bailey WC, Cohen SJ, et al. Smoking cessation. Clinical Practice Guideline No 18. Rockville, Maryland: US Department of Health and Human Services, Public Health Service, Agency for Health Care Policy and Research, April 1996. (AHCPR Publication No 96-0692).
- [Background] National Center for Health Statistics (US). Health, United States, 2004: With Chartbook on Trends in the Health of Americans. Hyattsville (MD): National Center for Health Statistics (US); 2004 Sep. Report No.: 2004-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK20751/ PMID 20698065
- [Background] Centers for Disease Control and Prevention (CDC). Tobacco use among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2006 Oct 27;55(42):1145-8. PMID 17065979
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 1994. MMWR Morb Mortal Wkly Rep. 1996 Jul 12;45(27):588-90. PMID 9132579
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2000. MMWR Morb Mortal Wkly Rep. 2002 Jul 26;51(29):642-5. PMID 12186222
- [Background] CDC. The Health Consequences of Smoking: Nicotine Addiction: A Report of the Surgeon General 1988. Rockville, MD: U.S. Department of Health and Human Services, CDC, Center for Health Promotion and Education, Office on Smoking and Health; 1988.
- [Background] CDC. Reducing Tobacco Use: A Report of the Surgeon General. Atlanta, GA: U.S. Department of Health and Human Services, CDC, Office on Smoking and Health; 2000.
- [Background] Fiore MC, Bailey WC, Cohen SJ, Dorfman SF, Goldstein MG, Gritz ER, et al. Treating Tobacco Use and Dependence: Quick Reference Guide for Clinicians. Rockville, MD: U.S. Department of Health and Human Services, Public Health Service; 2000.
- [Background] USDHHS. The health consequences of smoking: nicotine addiction. Rockville, Maryland: Office on Smoking and Health, 1988.
- [Background] Westman, E. C., Levin, E. D., & Rose, J. E. Smoking while wearing the nicotine patch: Is smoking satisfying or harmful? Clinical Research. 1992;40, 871A.
- [Background] Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Confirmatory validation of the Brief Questionnaire of Smoking Urges. Value in Health 2005;8(3):334.